CLINICAL TRIAL: NCT06778980
Title: Investigation of the Effect of Externally Vs. Internally Focused Techniques on Neck Region Muscle Activation During Postural Correction Exercises in Individuals with Forward Head Posture: Prospective Randomized Crossover Study
Brief Title: The Effect of Focus Approaches on Neck Region Muscle Activation
Acronym: EMG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, BEYZA YAZGAN DAĞLI, Research Assistant, Gazi University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BYDTEZ-2024/1; Gazi University (Other: Gazi University, Physiotherapy and Rehabilitation)
Record Dates: First submitted 2024-11-20; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Forward Head Posture
Keywords: muscle activation; external focus; internal focus; scapular retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- unguided scapular retraction (No Intervention): Participants will be asked to perform the scapular retraction exercise without any corrective cues for the cervical region.
- unguided prone T exercise (No Intervention): Participants will be asked to perform the prone T exercise without any corrective cues for the cervical region.
- scapular retraction exercise with External focus (Active Comparator): For external focus, participants will wear a headband with a laser light positioned on their forehead. The laser will be aligned to shine above and between the eyebrows. A flat wall will be placed in front of them, where the laser light is clearly visible. Participants will be instructed: "Bring your head into a chin tuck position and focus on the point where the laser hits the wall while performing the exercise."
  Interventions: Other: The chin tuck posture
- scapular retraction exercise with internal focus (Active Comparator): Participants will be instructed: "Bring your head into a chin tuck position and focus on keeping your neck in a neutral position while performing the exercise."
  Interventions: Other: The chin tuck posture
- prone T exercise with external focus (Active Comparator): For external focus, participants will wear a headband with a laser light positioned on their forehead. The laser will be aligned to shine above and between the eyebrows. A flat wall will be placed in front of them, where the laser light is clearly visible. Participants will be instructed: "Bring your head into a chin tuck position and focus on the point where the laser hits the wall while performing the exercise."
  Interventions: Other: The chin tuck posture
- prone T exercise with internal focus (Active Comparator): Participants will be instructed: "Bring your head into a chin tuck position and focus on keeping your neck in a neutral position while performing the exercise."
  Interventions: Other: The chin tuck posture

INTERVENTIONS:
Other: The chin tuck posture — A chin tuck is a posture correction technique where the individual gently tucks their chin towards their chest while keeping the rest of the body straight. This movement helps align the head and neck, reducing forward head posture and improving spinal alignment. After performing the unguided exercises, the patients will be taught the chin tuck position. From this point onward, they will be instructed to maintain the chin tuck position while performing the exercises using both external and internal focus strategies.
  Arms: prone T exercise with external focus; prone T exercise with internal focus; scapular retraction exercise with External focus; scapular retraction exercise with internal focus

SUMMARY:
Forward Head Posture (FHP) causes muscle imbalances in the neck and shoulder regions. Various exercises are suggested to correct FHP. During these exercises, internal and external focus techniques are used to enhance motor learning and improve muscle balance. However, there are no studies examining how these approaches affect neck muscle activation in individuals with FHP. Therefore, the purpose of this study is to investigate the effects of external and internal focus techniques, aimed at improving cervical alignment during postural correction exercises, on cervical muscle activation in individuals with FHP.

DETAILED DESCRIPTION:
Various corrective exercises are suggested in the literature to address Forward Head Posture (FHP). For individuals without musculoskeletal issues, chin-tuck and scapular retraction exercises in a supine position have strong evidence for effectiveness. Scapular stabilization exercises help reduce negative mechanical loads caused by abnormal scapular and cervical spine positions. Additionally, focusing attention on the exercise or target area is used to enhance motor learning and muscle balance, with external focus shown to improve performance in various tasks compared to internal focus.

In clinical practice, it is essential to maintain cervical alignment during scapular retraction exercises for individuals with FHP. To optimize muscle balance during these exercises, instructions often emphasize keeping the chin-tuck position to avoid cervical protraction. Internal and external focus approaches during scapular retraction exercises may help balance the muscle imbalances in individuals with FHP. However, no studies have yet examined the effects of internal and external focus approaches on neck muscle activation in individuals with FHP.

Thirty participants with FHP, defined as having a craniovertebral angle less than 50 degrees, will be included in the study. Participants will perform scapular retraction exercises (bilateral row) with a theraband and T-exercises in a prone position. The exercises will be carried out under three conditions: without guidance (control - no corrective cues for the cervical region), external focus, and internal focus. A laser headband will be used for the external focus condition. Muscle activation of the Upper Trapezius, Middle Trapezius, Lower Trapezius, Serratus Anterior, and Sternocleidomastoid muscles will be measured using the Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ). Muscle activation will be calculated as a percentage of Maximum Voluntary Isometric Contraction (MVIC), and the % MVIC values will be used for analysis. The order of exercises will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years,
* Craniovertebral angle (CVA) less than 50 degrees,
* Willing to not participate in any treatment/evaluation during the study,
* Voluntary participation.

Exclusion Criteria:

* Experiencing pain in the neck, spine, upper or lower extremities for the past 3 months,
* Body mass index (BMI) greater than 25 kg/m²,
* History of neck injuries or surgeries such as intervertebral disc herniation, spondylosis, radiculopathy, chronic headaches, or whiplash,
* Any visual, auditory, or sensory impairments,
* Temporomandibular joint issues,
* Neurological (e.g., epilepsy), rheumatological, or orthopedic symptoms,
* Any conditions affecting balance and muscle control,
* Cardiopulmonary or systemic diseases that prevent exercise.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-02 (Estimated); Primary Completion 2025-03-05 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) Measurement on neck muscles | through study completion, an average of 3 months
  The activation of the Upper Trapezius (UT), Middle Trapezius (MT), Lower Trapezius (LT), Serratus Anterior (SA), and Sternocleidomastoid (SCM) muscles will be measured using the non-invasive surface 8-channel EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ).
Craniovertebral Angle Measurement | through study completion, an average of 3 months
  The craniovertebral angle (CVA) will be measured using the reliable and valid lateral digital photogrammetric method and Kinovea Video Analysis Software. Participants will be filmed laterally from their dominant side (left for left-dominant, right for right-dominant). A phone on a tripod will be placed 1.5 meters away from the participant at shoulder height. Markers will be placed on the tragus and C7 spinous process for accurate measurement, with participants wearing tight shorts and a short-sleeved shirt. They will be instructed to stand with feet shoulder-width apart and face forward. Before photographing, participants will walk in place five times to capture their natural head-body position. Photos will be taken within the first 5 seconds, and the CVA will be measured using Kinovea Video Analysis Software.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No